CLINICAL TRIAL: NCT05480059
Title: Assessment of Psychological Symptoms and Health Related Quality of Life in Patients With Irritable Bowel Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Elhussiny Salah Mahmoud, Ahmed Elhussiny, Assiut University
Other Study IDs: Irritable bowel syndrome
Record Dates: First submitted 2022-07-28; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: IBS - Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: A questionnaire — A Questionnaire-based Assessment of the Psychiatric Co-morbidities and Health-related Quality of life in Patients with Irritable Bowel Syndrome

SUMMARY:
To evaluate the relation between the clinical presentations and the psychiatric co-morbidities with the quality of life in patients with irritable bowel syndrome.

DETAILED DESCRIPTION:
IBS is a chronic functional disorder characterized by abdominal pain and altered bowel habit in the absence of a specific and unique organic pathology.

Rome IV criteria is used to diagnose IBS patients which depends on the presence of recurrent abdominal pain on average at least 1 day per week in the last 3 months associated with 2 or more of the following; related to defecation, associated with change in frequency of stool , associated with change in stool form. These criteria should be fulfilled for the last 3 months with symptom onset at least 6 months before diagnosis.]1.[ brian et al 2017)[ IBS sub-types include 4 sub-types described according to the dominant stool pattern diarrhea (IBS -D) , constipation (IBS- C) , mixed ( IBS-M) , unspecified( IBS-U) subtypes . ] [2 Cristiane Kibune Nagasako et al 2016 [ The Identified Risk factors for IBS include female sex , younger age , psychological stress during or before infectious gastroenteritis , and the severity of enteritis. [3 ] Oh Young Lee et al 2010

IBS is a painful condition associated with significant psychological distress and psychiatric comorbidities such as higher levels of anxiety or depression and suicidal ideation, with a negative impact on quality of life [4 ] .Canavan et al., 2014; Stasiet al., 2014).

Major psychiatric disorders seen in patients were GAD and MDE. GAD was seen in 30.0% of patients having IBS while MDE was present in 28.0% [5]

Therefore, IBS consequences are measured in direct costs; medical treatment and procedures or indirect costs such as reduced productivit and low quality of life.[6] Doshi et al., 2014a However, few studies were conducted to evaluate the impact of clinical presentations or psychiatric co-morbidities with the quality of life in IBS.

ELIGIBILITY:
Inclusion Criteria:

* 1- Patient age between 18 - 50 years old 2- Patients fulfilling Rome IV criteria with normal investigations such as CBC, ESR , liver and kidney function and \ or colonoscopy 3- Healthy control: who do not fulfil Rome IV criteria with normal investigations

Exclusion Criteria:

* 1- Those older than 50 years of age with recent onset of symptoms (less than 6 months).

  2- Organic causes of colonic symptom. 3- Patients with IBS who have alarm signs. 4- Those with coexisting diseases (e.g. intestinal parasites, malignancy, diabetes mellitus cardiovascular pulmonary, hepatic, or renal disorder).

  5- Those with a family history of colorectal cancer. 6- IBS in children (< 18 years) and IBD-IBS patients

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Patient age between 18 - 50 years old, fulfilling Rome IV criteria with normal investigations
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Psychiatric Co-morbidities and Health-related Quality of life in Patients with Irritable Bowel Syndrome | baseline
  A Questionnaire-based Assessment of the Psychiatric Co-morbidities and Health-related Quality of life in Patients with Irritable Bowel Syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Ramadan, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lacy BE, Patel NK. Rome Criteria and a Diagnostic Approach to Irritable Bowel Syndrome. J Clin Med. 2017 Oct 26;6(11):99. doi: 10.3390/jcm6110099. PMID 29072609
- [Background] Kibune Nagasako C, Garcia Montes C, Silva Lorena SL, Mesquita MA. Irritable bowel syndrome subtypes: Clinical and psychological features, body mass index and comorbidities. Rev Esp Enferm Dig. 2016 Feb;108(2):59-64. doi: 10.17235/reed.2015.3979/2015. PMID 26838486
- [Background] Lee OY. Prevalence and risk factors of irritable bowel syndrome in Asia. J Neurogastroenterol Motil. 2010 Jan;16(1):5-7. doi: 10.5056/jnm.2010.16.1.5. Epub 2010 Jan 31. No abstract available. PMID 20535320